CLINICAL TRIAL: NCT03622307
Title: Subcutaneous ICD Therapy Combined With VT Ablation for the Secondary Prevention of Sudden Cardiac Death
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Eyal Nof, Dr. Eyal Nof Director Of Invasive Electrophysiology Service Davidai Arrhythmia Center Leviev Heart Center , Sheba Medical Center, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VT ablation/SICD study
Record Dates: First submitted 2018-06-05; First posted 2018-08-09 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Sudden Cardiac Death
Keywords: Subcutaneous ICD Therapy; VT Ablation
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- S-ICD therapy combined with VT Ablation (Experimental): To evaluate the feasibility and safety of a management approach that incorporates VT-ablation and S-ICD implantation in secondary prevention patients
  Interventions: Device: Subcutaneous ICD Therapy Combined with VT Ablation

INTERVENTIONS:
Device: Subcutaneous ICD Therapy Combined with VT Ablation — S-ICD implantation and VT ablation/substrate modification among patients with a secondary prevention indication for an ICD

SUMMARY:
This study evaluates the feasibility and safety of a management approach that incorporates VT-ablation and S-ICD implantation in secondary prevention patients. This is a single arm prospective study with 30 patients eligible for implantation of an ICD for the secondary prevention of sudden cardiac death.

DETAILED DESCRIPTION:
The subcutaneous ICD (S-ICD) is a system without transvenous leads that has been proven to safely provide defibrillation for patients at risk of sudden cardiac death due to ventricular tachyarrhythmias. However this system is currently not able to perform anti tachycardia pacing (ATP) which can terminate some VT, thus avoiding painful shocks.

Ideally slow VT should be managed with RF ablation while fast VT causing hemodynamic consequences should be treated with ICD shocks combined with medications. Typically, ICDs in secondary prevention patients are programmed to intervene at 10 msec at least above the clinical VT. In cases of hemodynamically stable VT this can result in unnecessary therapies and lead to ICD shocks. S-ICD can safely manage fast VTs while slower hemodynamically VTs can be managed with ablation.

This approach can avoid transvenous ICD related complications and unnecessary ICD interventions such as ATP which can accelerate VT to ICD shock zone. However, the benefit of this management strategy compared to conventional transvenous ICD programming has not been studied in patients who receive the device for the secondary prevention of sudden cardiac death.

ELIGIBILITY:
Inclusion Criteria:

* Any scar related sustained VT or VF
* Class I, IIa, or IIb indication for secondary prevention ICD therapy per ESC Guidelines
* Age ≥ 22 years on a date of consent
* LVEF ≤ 40%
* Positive ECG screening for S-ICD

Exclusion Criteria:

* A requirement for antibradycardia pacing or CRTD
* Subjects with an existing ICD, CRT, CRT-D, or pacemaker device.
* Contraindications for S-ICD implantation
* Contraindications for VT ablation
* Serious known concomitant disease with a life expectancy of < 1 year
* Elderly patients >80 years of age
* NYHA class IV or need for mechanical LV support (ECMO)
* Pregnancy or nursing
* Unwilling or unable to give informed consent

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
arrhythmic event | 24 months
  Occurrence of treated arrhythmic event (appropriate and inappropriate). The primary endpoint will be assessed by patient interview, clinical examination, and regularly scheduled SICD interrogation during follow-up

SECONDARY OUTCOMES:
Appropriate ICD therapy | 24 months
  Rate of appropriate ICD therapy (defined as a shock therapy for ventricular tachycardia or fibrillation).
  This will be assessed by patient interview and regularly scheduled ICD interrogation during follow-up.
Inappropriate ICD therapy | 24 months
  Rate of inappropriate therapy (defined as any ICD shock delivered for Non-VT event).
  This will be assessed by patient interview and regularly scheduled ICD interrogation during follow-up.
Ablation success rates | 24 months
  Rate of ablation success (defined as absence of Ventricular Arrhythmia). This will be assessed by patient interview and regularly scheduled ICD interrogation during follow-up.

OTHER OUTCOMES:
All cause mortality | 24 months
  Rate of all cause mortality. This will be assessed during patient follow up.
Cardiac mortality | 24 months
  Rate of all cardiac mortality. This will be assessed during patient follow up.